CLINICAL TRIAL: NCT04802616
Title: The Effect of Immunostimulation With Polyvalent Mechanical Bacterial Lysate on Changes in the Concentration of iNKT Cells in Children With Allergic Rhinitis.
Brief Title: The Influence of Nonspecific Immunostimulation on Changes in the Concentration of iNKT Cells
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Kamil Janeczek, Principal Investigator, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KE-0254/251/2020
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2021-08

CONDITIONS: Allergic Rhinitis Due to Grass Pollen
Keywords: allergic rhinitis; seasonal allergic rhinitis; children; grass pollen season; bacterial lysate; iNKT cells
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — Broncho-Vaxom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyvalent mechanical bacterial lysate (Experimental): Treatment over 3 successive months with one daily sublingual tablet (7 mg of bacterial lysate) over 10 days followed by 20 days of rest.
  Interventions: Drug: Ismigen
- Placebo (Placebo Comparator): Treatment over 3 successive months with one daily sublingual tablet over 10 days followed by 20 days of rest.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ismigen — Sublingual tablets containing 7 mg of bacterial lysate from the following bacteria: Staphylococcus aureus, Haemophilus influenzae serotype B, Klebsiella pneumoniae, Klebsiella ozaenae, Neiserria catarrhalis, Streptococcus viridans, Streptococcus pyogenes, Streptococcus pneumoniae (6 strains: TY1/EQ11, TY2/EQ22, TY3/EQ14, TY5/EQ15, TY8/EQ23, TY47/EQ24).
  Other Names: Polyvalent mechanical bacterial lysate (PMBL)
  Arms: Polyvalent mechanical bacterial lysate
Drug: Placebo — Matched tablets without any active substance.
  Arms: Placebo

SUMMARY:
The aim of the study is to assess the effect of polyvalent mechanical bacterial lysate (PMBL, Ismigen) on the clinical course of grass pollen-induced allergic rhinitis (using: total nasal symptom score, visual analogue scale, peak nasal inspiratory flow measurement) in children aged 5 to 17 and to assess changes in the concentration of iNKT cells under the influence of the therapy. Half of the 80 participants will receive PMBL while the other half will receive placebo.

DETAILED DESCRIPTION:
Seasonal allergic rhinitis (SAR) is caused by the allergens of wind-pollinated plants, and in Poland mainly by grass pollen allergens. During the grass pollen season, patients may suffer from fatigue, weakness, lack of fitness, difficulty in sleeping and reduced performance at school. In people allergic to the above-mentioned pollen, the disease significantly reduces the quality of life and requires intensive treatment in the pollen period.

Due to the high incidence of allergic rhinitis, the negative impact of the disease on the quality of life, and incomplete effectiveness of previously available therapeutic methods, new methods of treatment are being developed. Recent research highlights the immunoregulatory potential of bacterial lysates, indicating the possibility of their future use in the prevention and treatment of allergic diseases, including atopic dermatitis, allergic rhinitis, and asthma. However, the mechanism of action of these drugs in allergic diseases is still not entirely clear.

iNKT (Invariant Natural Killer T) are a conserved line of T cells with unique features expressing the invariant TCR alpha chain and recognizing glycolipids presented in the context of the non-classical MHC molecule, CD1d. As a result of TCR stimulation, iNKT cells are able to quickly secrete a variety of cytokines, thus stimulating various immune processes and playing an immunoregulatory role. iNKT cells are a small percentage of all T cells, however numerous studies indicate their possible participation in the pathogenesis of allergic diseases.The ambivalence of the activity of iNKT cells may result from the heterogeneity of this subpopulation. iNKT cells, like T lymphocytes, can be divided into further subpopulations: iNKT1, iNKT2, iNKT10, iNKT17 and iNKTreg. Individual subpopulations have a different cytokine profile, and thus may play opposite functions in the pathomechanism of many diseases, including allergic ones.

The main aim of this study is to evaluate the clinical course of the pollen allergic rhinitis, caused by grass pollen allergens in children during the grass pollen season, treated with polyvalent mechanical bacterial lysate (PMBL) and to assess the impact of PMBL on changes in the concentrations of the iNKT cell subpopulation. The approval of the Bioethics Committee at the Medical University in Lublin was obtained for the study.

Eighty children with SAR will be enrolled to this study and randomly assigned to the PMBL group (n=40) and placebo group (n=40). The study will include six visits, 2 site visits (before the grass pollen season and at the peak of the grass pollen season) and 4 telephone visits.The first site visit will be the randomization visit. The second site visit will take place after the end of the drug intake period. Telephone contact with the patient will take place twice during the period of taking the drug, and twice after the end of this period (follow-up visits).The time frame of the grass pollen season for south-eastern Poland will be determined using the "95%" method on the basis of measurements of grass pollen concentration in the atmospheric air, which will be obtained from the Environmental Allergy Research Centre in Warsaw. Patients will start taking sublingual tablets at the beginning of the April 2021.

Nasal SAR symptoms will be recorded by parents of children in the daily patient diary according to the standard scoring system (TNSS, total nasal symptom score), and their intensity will be also evaluated during six visits using VAS (visual analogue scale). At each site visit, peak nasal inspiratory flow (PNIF) will be also measured.

In order to determine the mechanism responsible for the possible effects of PMBL, blood samples (8 ml) will be taken from patients for additional tests during two site visits. The following iNKT cell subpopulations will be measured in the blood: iNKT1, iNKT2, iNKT10, iNKT17 and iNKTreg.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders aged 5 to 17 years.
* Children with grass pollen-induced allergic rhinitis recognized and treated according to current ARIA (Allergic Rhinitis and its Impact on Asthma) recommendations.
* Positive skin prick test to grass pollen allergens or positive specific IgE (defined as ≥ class 2, ≥ 0,70 kU/l) against timothy grass pollen allergens.
* Presentation of clinical symptoms of the allergic rhinitis (rhinorrhea, nasal congestion, nasal itching, sneezing) in at least two recent grass pollen seasons in Poland before inclusion in the study.
* Proper use of polyvalent mechanical bacterial lysate sublingual tablets.
* Not using drugs to alleviate the symptoms of allergic rhinitis in the last 7 days prior to enrollment in the study: intranasal glucocorticosteroids, intranasal, oral and ophthalmic antihistamines, intranasal and oral alpha-mimetics, intranasal anticholinergics, antileukotrienes and cromones.
* Written informed consent obtained from parents/guardians before any study related procedures are performed.

Exclusion Criteria:

* Patient received mechanical bacterial lysate immunostimulation within the previous 12 months before randomisation visit.
* Patient received chemical bacterial lysate immunostimulation within the previous 6 months before randomisation visit.
* Patient received oral/subcutaneous allergen-immunotherapy within the previous 3 years before the start of the study.
* Other chronic conditions of the nose or nasal sinuses.
* Severe nasal septum deviation.
* Acute respiratory infection in the 2 weeks prior to randomization visit.
* Treatment with systemic corticosteroids within the last 6 months before the start of the study.
* History of transfusion of blood, blood components or blood products.
* Pregnant or breastfeeding woman.
* Other chronic, uncontrolled diseases of the respiratory tract, gastrointestinal tract, urinary system, hematological diseases, immunodeficiency, cancer, cystic fibrosis.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Change in the severity of nasal SAR symptoms as assessed by total nasal symptom score (TNSS) | at baseline, at 1-month, at 2-months, at 3-months, at 4-months and at 5-months
  The severity of nasal SAR symptoms (sneezing, runny nose, itchy nose and nasal congestion) will be recorded by parents of children in the daily patient diary using the following scale: 0 = absent (no symptom); 1 = mild (symptom present, easily tolerated); 2 = moderate (awareness of symptom, bothersome but tolerable); 3 = severe (symptoms hard to tolerate, interfere with daily activities and/or sleeping).
  The total nasal symptom score (sum of the 4 symptom scores) ranges from 0 (no symptoms) to 12 (worst symptoms).
  Weekly average TNSS values from the baseline period (before the grass pollen season) and obtained 1 month, 2 months, 3 months, 4 months and 5 months after initiating therapy will be used for statistical analysis.
Change in the nasal obstruction using peak nasal inspiratory flow (PNIF) | at baseline and at 3-months
  Assessment of the nasal obstruction during two site visits based on measurement of peak nasal inspiratory flow by Youlten Peak Flow Meter (Clement Clarke International, UK).
  The higher PNIF value, the smaller nasal obstruction.
Change in the severity of nasal SAR symptoms as assessed by visual analogue scale (VAS) | at baseline, at 1-month, at 2-months, at 3-months, at 4-months and at 5-months
  Assessment of the severity of nasal SAR symptoms during six visits (2 site visits and 4 telephone visits) with the use of visual analogue scale.The patient will be asked to indicate the severity of nasal SAR symptoms on a 100 mm visual analogue scale, where 0 is no symptoms and 100 the worst possible symptoms.
iNKT1 cells concentration | at baseline and at 3-months
  To assess the change in the level of iNKT1 cells (T-bet+IFN-γ+) in the blood.
iNKT2 cells concentration | at baseline and at 3-months
  To assess the change in the level of iNKT2 cells (GATA3+IL-4+) in the blood.
iNKT10 cells concentration | at baseline and at 3-months
  To assess the change in the level of iNKT10 cells (E4BP4+IL-10+) in the blood.
iNKT17 cells concentration | at baseline and at 3-months
  To assess the change in the level of iNKT17 cells (RORγt+IL-17+) in the blood.
iNKTreg cells concentration | at baseline and at 3-months
  To assess the change in the level of iNKTreg cells (FoxP3+) in the blood.

SECONDARY OUTCOMES:
Frequency of oral H1-antihistamines use | from baseline, up to the 5-month time point
  To assess the mean number of days of oral H1-antihistamines use for the relief of SAR symptoms.
Frequency of intranasal corticosteroids use | from baseline, up to the 5-month time point
  To assess the mean number of days of intranasal corticosteroids use for the relief of SAR symptoms.
Incidence of treatment emergent adverse events [safety and tolerability] | from baseline, up to the 5-month time point
  Incidence, frequency and severity of treatment emergent adverse events.
Incidence of treatment emergent adverse events leading to discontinuation [safety and tolerability] | from baseline, up to the 5-month time point
  The number of participants with adverse events leading to discontinuation.
Time to discontinuation due to treatment emergent adverse events [safety and tolerability] | From date of randomization until the date of occurrence of an adverse event leading to discontinuation, assessed up to 5 months
  To assess the time that has elapsed since treatment initiation to the occurrence of an adverse event leading to discontinuation.
Incidence of treatment emergent abnormalities in physical examination findings [safety and tolerability] | at baseline and at 3-months
  Observe skin, lymph nodes, ears, eyes, nose, throat, cardiac and pulmonary status, abdomen and extremities for any abnormalities.
Incidence of treatment emergent abnormalities in pulse rate [safety and tolerability] | at baseline and at 3-months
  Measure resting pulse rate as beats per minute.
Incidence of treatment emergent abnormalities in blood pressure [safety and tolerability] | at baseline and at 3-months
  Measure systolic and diastolic blood pressure (in mmHg).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary Diseases and Children Rheumatology, Medical University of Lublin, Lublin, Poland

REFERENCES:
- [Background] Janeczek K, Emeryk A, Rachel M, Duma D, Zimmer L, Poleszak E. Polyvalent Mechanical Bacterial Lysate Administration Improves the Clinical Course of Grass Pollen-Induced Allergic Rhinitis in Children: A Randomized Controlled Trial. J Allergy Clin Immunol Pract. 2021 Jan;9(1):453-462. doi: 10.1016/j.jaip.2020.08.025. Epub 2020 Aug 26. PMID 32858239
- [Background] Janeczek KP, Emeryk A, Rapiejko P. Effect of polyvalent bacterial lysate on the clinical course of pollen allergic rhinitis in children. Postepy Dermatol Alergol. 2019 Aug;36(4):504-505. doi: 10.5114/ada.2019.87457. Epub 2019 Aug 30. No abstract available. PMID 31616231
- [Background] Banche G, Allizond V, Mandras N, Garzaro M, Cavallo GP, Baldi C, Scutera S, Musso T, Roana J, Tullio V, Carlone NA, Cuffini AM. Improvement of clinical response in allergic rhinitis patients treated with an oral immunostimulating bacterial lysate: in vivo immunological effects. Int J Immunopathol Pharmacol. 2007 Jan-Mar;20(1):129-38. doi: 10.1177/039463200702000115. PMID 17346436
- [Background] Meng Q, Li P, Li Y, Chen J, Wang L, He L, Xie J, Gao X. Broncho-vaxom alleviates persistent allergic rhinitis in patients by improving Th1/Th2 cytokine balance of nasal mucosa. Rhinology. 2019 Dec 1;57(6):451-459. doi: 10.4193/Rhin19.161. PMID 31403136
- [Background] Han L, Zheng CP, Sun YQ, Xu G, Wen W, Fu QL. A bacterial extract of OM-85 Broncho-Vaxom prevents allergic rhinitis in mice. Am J Rhinol Allergy. 2014 Mar-Apr;28(2):110-6. doi: 10.2500/ajra.2013.27.4021. PMID 24717947
- [Background] Liu C, Huang R, Yao R, Yang A. The Immunotherapeutic Role of Bacterial Lysates in a Mouse Model of Asthma. Lung. 2017 Oct;195(5):563-569. doi: 10.1007/s00408-017-0003-8. Epub 2017 May 4. PMID 28474108
- [Background] Esposito S, Soto-Martinez ME, Feleszko W, Jones MH, Shen KL, Schaad UB. Nonspecific immunomodulators for recurrent respiratory tract infections, wheezing and asthma in children: a systematic review of mechanistic and clinical evidence. Curr Opin Allergy Clin Immunol. 2018 Jun;18(3):198-209. doi: 10.1097/ACI.0000000000000433. PMID 29561355
- [Background] Emeryk A, Bartkowiak-Emeryk M, Raus Z, Braido F, Ferlazzo G, Melioli G. Mechanical bacterial lysate administration prevents exacerbation in allergic asthmatic children-The EOLIA study. Pediatr Allergy Immunol. 2018 Jun;29(4):394-401. doi: 10.1111/pai.12894. PMID 29575037
- [Background] Kronenberg M. Toward an understanding of NKT cell biology: progress and paradoxes. Annu Rev Immunol. 2005;23:877-900. doi: 10.1146/annurev.immunol.23.021704.115742. PMID 15771592
- [Background] Carnaud C, Lee D, Donnars O, Park SH, Beavis A, Koezuka Y, Bendelac A. Cutting edge: Cross-talk between cells of the innate immune system: NKT cells rapidly activate NK cells. J Immunol. 1999 Nov 1;163(9):4647-50. PMID 10528160
- [Background] Oki S, Miyake S. Invariant natural killer T (iNKT) cells in asthma: a novel insight into the pathogenesis of asthma and the therapeutic implication of glycolipid ligands for allergic diseases. Allergol Int. 2007 Mar;56(1):7-14. doi: 10.2332/allergolint.R-06-137. Epub 2007 Jan 29. PMID 17259804
- [Background] Bennstein SB. Unraveling Natural Killer T-Cells Development. Front Immunol. 2018 Jan 9;8:1950. doi: 10.3389/fimmu.2017.01950. eCollection 2017. PMID 29375573
- [Background] Gupta RK, Gupta K, Dwivedi PD. Pathophysiology of IL-33 and IL-17 in allergic disorders. Cytokine Growth Factor Rev. 2017 Dec;38:22-36. doi: 10.1016/j.cytogfr.2017.09.005. Epub 2017 Nov 11. PMID 29153708
- [Background] Coomes SM, Kannan Y, Pelly VS, Entwistle LJ, Guidi R, Perez-Lloret J, Nikolov N, Muller W, Wilson MS. CD4+ Th2 cells are directly regulated by IL-10 during allergic airway inflammation. Mucosal Immunol. 2017 Jan;10(1):150-161. doi: 10.1038/mi.2016.47. Epub 2016 May 11. PMID 27166557
- [Derived] Janeczek K, Kowalska W, Zarobkiewicz M, Suszczyk D, Mikolajczyk M, Markut-Miotla E, Morawska-Michalska I, Bakiera A, Tomczak A, Kaczynska A, Emeryk A, Rolinski J, Piotrowska-Weryszko K. Effect of immunostimulation with bacterial lysate on the clinical course of allergic rhinitis and the level of gammadeltaT, iNKT and cytotoxic T cells in children sensitized to grass pollen allergens: A randomized controlled trial. Front Immunol. 2023 Jan 17;14:1073788. doi: 10.3389/fimmu.2023.1073788. eCollection 2023. PMID 36733480